CLINICAL TRIAL: NCT06509594
Title: Effects of Scapular Stabilization Exercises Versus Eccentric Muscle Energy Techniques on Pain, Functional Disability and Postural Alignment in Patients With Upper Crossed Syndrome
Brief Title: Scapular Stabilization Exercises Versus Eccentric Muscle Energy Techniques in Patients With Upper Crossed Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/01111
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Upper Crossed Syndrome
Keywords: Upper Crossed Syndrome, Scapular Stabilization Exercises, Eccentric Muscle Energy technique, Pain, Functional disability
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A will be treated with Scapular Stabilization Exercises along with hot pack; (Active Comparator): Participants in the exercise group performed three scapular stabilization exercises at 3 sets of 10 repetitions, holding 10 seconds per one repetition, 5 days per week for 4 weeks under supervision. The exercises included:
  Interventions: Other: Protocol of Scapular Stabilization Exercises;
- Group B will be treated with Eccentric Muscle Energy Technique along with hot pack. (Active Comparator): Eccentric muscle energy technique was applied to subjects' cervical spine. The Cervical spine was brought to the barrier of motion in each plane i.e. Flexion/extension, lateral bending and rotation. Then subjects were asked to push their heads into the direction opposite that of the barrier. The therapist provided Isometric resistance for 7-10 seconds, after which the subjects relaxed their muscles completely and the therapist applied stretch. Three to five repetitions were performed(2). We will apply protocol for 4 weeks 20 Sessions (5 sessions in a week) and 10 sec rest between each segment with 3-5 time's repetition than their will 7-10 sec Isometric contraction followed by 5 sec relaxation than 30 sec hold for MET stretch.
  Interventions: Other: Protocol of Muscle Energy technique;

INTERVENTIONS:
Other: Protocol of Scapular Stabilization Exercises; — Exercise for the middle trapezius and rhomboid muscles: Participants were instructed to stand with their arms hanging beside their bodies. Then, they were instructed to flex their elbows 90◦ holding an elastic band and performing an external rotation of the shoulder, pulling both scapula together. Subsequently, they returned to a neutral shoulder position with elbow flexion.
  Exercise for the lower trapezius muscle: Participants were instructed to lie down in a prone position while holding an elastic band attached at one end under a mattress. They were then instructed to raise their shoulder 140◦.
  Exercise for the serratus anterior muscle: Participants were instructed to stand and flex their elbows 90◦ while holding an elastic band fixed behind the participants. Next, they were instructed to move the arm forward with a protracted scapula.
  Arms: Group A will be treated with Scapular Stabilization Exercises along with hot pack;
Other: Protocol of Muscle Energy technique; — During upper trapezius stretching, the participants were in seated position by holding the chair with one arm, and laterally tilted the head to the opposite side with the other hand pushing the head to increase lateral stretch.
  For pectoralis muscle stretch, participants were asked to stand in front of the Doorframe with elbow bent at 90 degree and was asked to lean forward without Taking a step forward. The stretch is felt across the anterior chest, which is held for 15-30 seconds with 2-3 repetitions. For levator scapulae stretch, the subjects were asked to take the seated position while holding the chair with one hand in order to maintain shoulder depression, then To flex and rotate neck to the opposite side by placing the other hand at the back of their head and to slowly pull it down toward the armpit.
  Arms: Group B will be treated with Eccentric Muscle Energy Technique along with hot pack.

SUMMARY:
This study will be a Randomized Clinical Trial in which Scapular Stabilization Exercises and Eccentric Muscle Energy technique will be applied on the individuals with upper crossed syndrome and changes will be recorded using different method and tools. Convenient sampling technique will be used to collect the data. The sample size of 34 patients will be recruited. Patients will be randomly allocated into two different groups through sealed envelope method. 17 patients will be allocated in each group. Group A will be treated with Scapular Stabilization Exercises along with hot pack; Group B will be treated with Eccentric Muscle Energy Technique along with hot pack. Craniovertebral Angle (CVA), Numeric Pain Rating Scale (NPRS), and Neck Disability Index (NDI) will be used as Data collecting tools.

DETAILED DESCRIPTION:
Upper Crossed Syndrome is defined byJanda as the involvement of different muscles of skeletal system which leads to shortness and tightness of anterior and upper trunk or weakness of posterior part of skeletal muscles. Alteration of muscles activity such as facilitation of different muscles as levator scapula, sternocleidomastoid, pectoralis muscles and inhibition of cervical flexors, serratus anterior The muscular imbalance occurs because of weak/tight and tonic muscles. Neck pain is the most frequent problem in developed countries. The prevalence of neck pain is approximately 10-15%. Neck pain is the most common reason for patients visiting healthcare professionals. Poor posture typically causes upper cross syndrome (UCS), resulting in neck pain. This syndrome can cause dysfunctional tone in posture and muscular disparity of head, neck and shoulder region.

ELIGIBILITY:
Inclusion Criteria:

* • Age: participants having range 18-35 years both male and female are included.

  * Craniovertebral angle<52
  * NPRS>3 and NDI>10
  * Patients having neck pain during movements.
  * Patients having neck pain due to sustained posture and after activity

Exclusion Criteria:

* Inflammation malignancy, neurological disorder
* Metabolic disorders
* Neck pain radiating into arms and upper extremity
* Neck pain associated with headache and facial pain
* Recent surgery
* History of recent trauma and fractures of cervical spine
* Patients having any other therapeutic intervention or medical treatment.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 4 weeks
  The NPRS was used to capture the patient's level of pain. Patients were asked to indicate the intensity of their current pain level using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable)(8).
  0 = no pain
  1 to 4 indicate mild pain 5 or 6 indicate moderate pain 7 to 10 indicate severe pain NPRS exhibited moderate reliability (ICC = 0.67) in t

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | 4 weeks
  The NDI consists of ten items. Each item has six different assertions expressing progressive levels of pain or limitation in activities. Item scores range from 0 (no pain or limitation) to 5 (as much pain as possible or maximal limitation). The total NDI score ranges from 0 to 5 points.

OTHER OUTCOMES:
Photogrammetry | 4 weeks
  A digital imaging technique will be used to evaluate head and neck posture in the standing position.

CONTACTS AND LOCATIONS:
Overall Officials: Dr hajira Anwer, M.S, Principal Investigator — Riphah International University
Locations (1):
- Faisal masaood teaching hospital Sargodha, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salahzadeh Z, Maroufi N, Ahmadi A, Behtash H, Razmjoo A, Gohari M, Parnianpour M. Assessment of forward head posture in females: observational and photogrammetry methods. J Back Musculoskelet Rehabil. 2014;27(2):131-9. doi: 10.3233/BMR-130426. PMID 23963268
- [Background] Gillani SN, Ain Q-, Rehman SU, Masood T. Effects of eccentric muscle energy technique versus static stretching exercises in the management of cervical dysfunction in upper cross syndrome: a randomized control trial. J Pak Med Assoc. 2020 Mar;70(3):394-398. doi: 10.5455/JPMA.300417. PMID 32207413
- [Background] Kang JI, Choi HH, Jeong DK, Choi H, Moon YJ, Park JS. Effect of scapular stabilization exercise on neck alignment and muscle activity in patients with forward head posture. J Phys Ther Sci. 2018 Jun;30(6):804-808. doi: 10.1589/jpts.30.804. Epub 2018 Jun 12. PMID 29950768
- [Background] Ali S, Ahmad S, Jalal Y, Shah B. Effectiveness of Stretching Exercises Versus Muscle Energy Techniques in the Management of Upper Cross Syndrome: JRCRS. 2017; 5 (1): 12-16. Journal Riphah College of Rehabilitation Sciences. 2017;5(1):12-6.
- [Background] Sasidharan S. Comparing the effectiveness of muscle energy technique and static stretching in upper crossed syndrome on IT professionals: City University.
- [Background] IBRAHIM ME, HANAN SE-S, ABDELSALAM S. Cervical Stabilization Exercises Versus Scapular Stabilization Exercises in Treatment of Chronic Mechanical Neck Pain. The Medical Journal of Cairo University. 2022;90(9):1729-35.
- [Background] Sakshi N, Suman M, Geetanjali S. Effect of muscle energy technique and deep neck flexors exercise on pain, disability and forward head posture in patients with chronic neck pain. National Editorial Advisory Board. 2014;8(4):43.
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Background] Jorritsma W, Dijkstra PU, de Vries GE, Geertzen JH, Reneman MF. Detecting relevant changes and responsiveness of Neck Pain and Disability Scale and Neck Disability Index. Eur Spine J. 2012 Dec;21(12):2550-7. doi: 10.1007/s00586-012-2407-8. Epub 2012 Jul 3. PMID 22752592
- [Background] Nitayarak H, Charntaraviroj P. Effects of scapular stabilization exercises on posture and muscle imbalances in women with upper crossed syndrome: A randomized controlled trial. J Back Musculoskelet Rehabil. 2021;34(6):1031-1040. doi: 10.3233/BMR-200088. PMID 34151819